CLINICAL TRIAL: NCT01037075
Title: Influence of Nicotine on Cognitive Function in Schizophrenic Patients With and Without Comorbid Drug Dependence
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Maryland, College Park (Other)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906400; 06-DA-N400; NCT00686153 (obsolete NCT alias)
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2013-01-22

CONDITIONS: Schizophrenia; Drug Abuse/Dependency
Keywords: Schizophrenia; Dual Diagnosis; Nicotine Nasal Spray; Drug Abuse/Dependence; Cognitive Processes
MeSH Terms: conditions — Schizophrenia; Substance-Related Disorders

SUMMARY:
Background:

* Individuals with schizophrenia have a significantly higher tendency to develop substance abuse or dependence than the general population. For instance, people with schizophrenia smoke much more than the general population, and many are dependent on street drugs such as cocaine and heroin. However, these individuals are rarely included in research studies that might provide more information about treatments for both schizophrenia and substance abuse.
* Strong evidence suggests that schizophrenia and substance dependence have similar effects on the brain, affecting attention, memory, and eye movement. Other research indicates that schizophrenia and substance dependence affect the same parts of the dopamine system, contributing to problems in brain function that require treatment. These new developments provide a strong rationale to study the combination of schizophrenia and substance dependence.
* Nicotine may help improve brain function and thinking in individuals with both schizophrenia and drug dependence. Some of the thinking and memory problems experienced by these individuals can be treated with nicotine. However, more research is needed to determine exactly how nicotine affects individuals with both schizophrenia and drug dependence.

Objectives:

* To determine whether individuals with schizophrenia and drug dependence show impairment in tests of eye tracking, attention, and memory compared with healthy control subjects.
* To evaluate the effect of nicotine on eye tracking, attention, and memory in individuals with both schizophrenia and substance dependence.

Eligibility:

- Current smokers (at least 10 cigarettes per day for the past year) between 18 and 55 years of age who (1) have been diagnosed with schizophrenia/schizoaffective disorder, (2) have been diagnosed with schizophrenia/schizoaffective disorder and are currently using heroin and/or cocaine, or (3) are healthy individuals with no family history of psychotic illness.

Design:

* The study will consist of one training session and three testing sessions. Each session will last about 2 hours.
* The training session will introduce participants to the study tests and evaluate their tolerance of the nicotine nasal spray used in the study. Participants who cannot tolerate the higher dose of the spray will not continue in the study.
* At the start of each testing session, smokers will have one cigarette to standardize the time of the most recent exposure to nicotine.
* During the testing sessions, participants will receive a placebo spray, a lower dose of nicotine, or a higher dose of nicotine, and then will be asked to perform tests that evaluate attention, memory, and other thinking tasks.

DETAILED DESCRIPTION:
Objective:

Specific aim 1: To test the hypothesis that individuals with comorbid schizophrenia and drug dependence will show impaired neurocognitive functions in anticipatory learning of eyetracking, attention, and memory performance compared to healthy controls subjects.

Specific aim 2: To test the hypothesis that nicotine will dose-dependently improve anticipatory learning of eyetracking, attention, and memory performance in individuals with comorbid schizophrenia and substance dependence.

Study Population:

Male and nonpregnant-female smokers 18 to 55 years of age, from the following subject groups: (1) patients with a DSM IV diagnosis of schizophrenia (2) patients with dual DSM IV diagnoses of schizophrenia and heroin and/or cocaine dependence or abuse, or on methadone or beprenorphine maintenance and (3) healthy individuals with no family history of psychotic illness.

Design:

This study will be a double-blind, placebo controlled trial of nicotine or placebo nasal sprays. Participants will have four visits. After the training session, participants will be administered one dose (0, 1 or 2 mg) of nicotine nasal spray during each of the 3 experimental sessions. The dose will be given 5 minutes prior to the cognitive task batteries.

Outcome Measures:

Vital signs, moods, and performance on tasks assessing eye movement (initiation latency, initiation acceleration, closed-loop pursuit gain), attention (Continuous Performance and Digit Symbol Substitution Tasks), and memory (delayed recognition and nback).

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants must meet the following criteria:

* age 18 60
* smoke 10 or more cigarettes/day for at least the past year

Experimental groups 1 and 2, additional criteria:

-DSM-IV diagnosis of schizophrenia or schizoaffective disorder (assessments pertaining to these diagnoses will be done in other MPRC screening protocols).

Experimental group 2, additional criteria:

-DSM-IV diagnosis of abuse or dependence on cocaine and/or heroin or on methadone or buprenorphine maintenance.

EXCLUSION CRITERIA:

Comprehensive medical history:

-Exclusions: Heart disease, uncontrolled blood pressure (persistent systolic above 155 or diastolic above 95), neurological conditions (stroke, seizure, history of head injury), asthma, emphysema, chronic bronchitis, chronic obstructive pulmonary disease, pathology of nasal passages that precludes the effective administration of nicotine nasal spray.

Drug Use Survey

All subjects:

* Exclude if treatment for tobacco dependence during the previous 6 months.
* Healthy controls and schizophrenic patients without comorbid drug abuse or dependence: Exclude if history alcohol or other substance dependence ever, or alcohol or other substance abuse in the past year. Verify abstinence from controlled substances with urine screen (Iscreen). Participants in the above 2 groups who are positive for any illicit drug (with the exception of marijuana) will be excluded.

Structured Clinical Interview for DSM-IV

-Healthy controls: exclude if any current psychiatric disorder

Urine pregnancy for females:

-Exclude if positive.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2006-05-14; Study Completion 2013-01-22

CONTACTS AND LOCATIONS:
Overall Officials: Carol Myers, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (2):
- United States (2):
  - National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland
  - Matthews Media Group, Rockville, Maryland

REFERENCES:
- [Background] Avila MT, Sherr JD, Hong E, Myers CS, Thaker GK. Effects of nicotine on leading saccades during smooth pursuit eye movements in smokers and nonsmokers with schizophrenia. Neuropsychopharmacology. 2003 Dec;28(12):2184-91. doi: 10.1038/sj.npp.1300265. PMID 12968127
- [Background] Bennett ME, Bellack AS, Gearon JS. Treating substance abuse in schizophrenia. An initial report. J Subst Abuse Treat. 2001 Mar;20(2):163-75. doi: 10.1016/s0740-5472(00)00167-7. PMID 11306219
- [Background] Berman SM, Martinez RA, Noble EP. Familial alcoholism and ERPs: differences in probability sensitivity? Alcohol Alcohol. 1993 Nov;28(6):695-707. PMID 8147978